CLINICAL TRIAL: NCT05847439
Title: A Phase 1, Single-center, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]BMS-986419 in Healthy Male Participants
Brief Title: A Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]BMS-986419 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN007-1004
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Metabolite profile; Radioactivity; BMS-986419; Healthy volunteer; Healthy participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]BMS-986419 (Experimental)
  Interventions: Drug: [14C]BMS-986419

INTERVENTIONS:
Drug: [14C]BMS-986419 — Specified dose on specified days
  Other Names: BMS-986419; EOAI4018683

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), metabolite profile, routes and extent of elimination, mass balance, as well as safety and tolerability of [14C]BMS-986419 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 33.0 kilograms/meter square (kg/m^2), inclusive, at screening. Body mass index = weight (kg)/(height [m])2.
* Healthy male participants as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [for example, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in (Day -2).

Exclusion Criteria:

* Any significant acute or chronic medical conditions.
* Any major surgery within 30 days of study intervention administration, such as gastrointestinal surgery (for example, cholecystectomy and any other gastrointestinal surgery) that could impact the absorption of study intervention (uncomplicated appendectomy and hernia repair are acceptable).
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease that could impact the absorption of study treatment.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 20
Time of maximum plasma observed concentration (Tmax) | Up to Day 20
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Up to Day 20
Total radioactivity recovered in urine (UR) | Up to Day 30
Total radioactivity recovered in feces (FR) | Up to Day 30
Total radioactivity recovered in bile (BR) | Up to Day 30
Total radioactivity recovered (Rtotal) | Up to Day 30
Percent of total radioactivity recovered (%Total) | Up to Day 30
Percent of total radioactivity recovered in urine (%UR) | Up to Day 30
Percent of total radioactivity recovered in feces (%FR) | Up to Day 30

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 60
Number of Participants with Serious AEs (SAEs) | Up to Day 60
Number of Participants with AEs leading to discontinuation | Up to Day 60
Number of Participants with Vital Sign Abnormalities | Up to Day 30
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 30
Number of Participants with Physical Examination Abnormalities | Up to Day 30
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Labcorp Clinical Research Unit - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome